CLINICAL TRIAL: NCT01315145
Title: MiDAS III (Mild® Decompression Alternative to Open Surgery): Vertos Mild Patient Evaluation Study
Acronym: MiDAS III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vertos Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MiDAS III
Record Dates: First submitted 2011-03-11; First posted 2011-03-15 (Estimated); Results first posted 2015-08-19 (Estimated); Last update posted 2015-08-31 (Estimated); Status verified 2015-08

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Percutaneous Lumbar Decompression (Active Comparator): Patients receiving percutaneous decompression using the mild® Device Kit.
  Interventions: Procedure: Percutaneous Lumbar Decompression
- Lumbar Epidural Steroid Injection (Active Comparator): Injection of epidural steroids into the lumbar spine
  Interventions: Drug: Epidural Steroid Injection

INTERVENTIONS:
Procedure: Percutaneous Lumbar Decompression — The percutaneous procedure is performed under fluoroscopic guidance to effect a lumbar decompression with minimal surrounding tissue and bone disruption. The mild® Device Kit is utilized to access, capture and remove bone and tissue.
  Other Names: mild procedure; mild lumbar decompression
  Arms: Percutaneous Lumbar Decompression
Drug: Epidural Steroid Injection — Injection of epidural steroids into the lumbar spine
  Other Names: ESI
  Arms: Lumbar Epidural Steroid Injection

SUMMARY:
This is a multi-center, prospective, observational clinical study to compare patient outcomes following treatment with either the mild® procedure or epidural steroid injection in patients with moderate to severe lumbar spinal stenosis exhibiting neurogenic claudication.

DETAILED DESCRIPTION:
The study was initially designed as a randomized trial. Due to difficulty of enrollment, the study was amended and converted to an observational comparative study with study arm being self-selected by the patient.

ELIGIBILITY:
Inclusion Criteria:

* Lumbar spinal stenosis (LSS) with neurogenic claudication where the Visual Analog Scale (VAS) of back and leg pain average is ≥ 5.
* Prior failure of conservative therapy.
* Oswestry Disability Index (ODI) score of ≥ 31%.
* Radiologic evidence of LSS, with unilateral or bilateral ligamentum flavum ≥ 4.1mm confirmed by pre-op MRI performed within 6-12 months of baseline visit.
* Able to walk ≥ 10 feet before being limited by pain.
* Available to complete 24-months of follow-up.
* Adults ≥ 50 years of age.

Exclusion Criteria:

* Prior surgery at intended treatment level.
* History of spinal fractures with current related pain symptoms.
* Motor deficit or disabling back and/or leg pain from causes other than LSS neurogenic claudication (e.g. acute compression fracture, metabolic neuropathy, vascular claudication symptoms, etc.).
* Significant/symptomatic disc protrusion or osteophyte formation judged by the Investigator as possible confounding factor to study results.
* Excessive facet hypertrophy judged by the Investigator as possible confounding factor to study results.
* Significant symptomatic foraminal stenosis.
* Confirmed anterior or retro-listhesis ≥ 3mm.
* Bleeding disorders and/or current use of anti-coagulants with the inability to withhold anticoagulants for required time prior to procedure.
* Able to walk ≥ 200 yards unaided in erect non-flexed position before being limited by pain.
* Able to stand ≥ 15 minutes in erect, non-flexed position before being limited by pain.
* Use of acetylsalicylic acid (ASA) and/or non-steroidal anti-inflammatory drug (NSAID) within 7 days of treatment.
* Pregnant and/or breastfeeding.
* Body mass index (BMI) ≥ 32 as calculated using the patient's weight multiplied by 703 then divided by height in inches squared.
* Epidural steroid, systemic steroid or any spine interventional procedure within prior six weeks of study procedure.
* Dementia and/or inability to give informed consent and to understand and complete follow-up patient reported outcomes forms.
* Inability of the patient to lie prone for any reason with anesthesia support (e.g. chronic obstructive pulmonary disease (COPD), obesity, etc.).
* On (or pending) Workman's Compensation or known to be considering litigation associated with back pain.
* Unable to tolerate MRI (pacemaker, spinal cord stimulator, etc.).
* Intrathecal pump.
* Any medical condition determined by the Investigator that would not allow subject to fulfill trial requirements or safely tolerate procedures in this study.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2011-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nagy Mekhail, MD, Principal Investigator — The Cleveland Clinic
Locations (27):
- United States (27):
  - HOPE Research Institute, Phoenix, Arizona
  - Center for Pain and Supportive Care, Scottsdale, Arizona
  - Pain Clinic of Monterey Bay, Aptos, California
  - Pain Control Associates of San Diego, Chula Vista, California
  - Navarro Pain Control Group, Inc., Solana Beach, California
  - IPM Medical Group, Inc., Walnut Creek, California
  - The GW Pain Center, Washington D.C., District of Columbia
  - Interventional Pain Physicians of South Florida, Aventura, Florida
  - Coastal Orthopedics and Sports Medicine, Bradenton, Florida
  - Holy Cross Interventional Spine & Pain Medicine Center, Fort Lauderdale, Florida
  - Space Coast Pain Institute, Merritt Island, Florida
  - Millennium Pain Center, Bloomington, Illinois
  - Commonwealth Pain Specialists, PLLC, Frankfort, Kentucky
  - The Spine Center Baltimore, Baltimore, Maryland
  - Michigan Pain Specialists, Ann Arbor, Michigan
  - Michigan Interventional Pain Center, Brownstown Twp., Michigan
  - Occupational and Pain Management Professionals, Crystal City, Missouri
  - Lab2Marche' LLC, Las Vegas, Nevada
  - Virtua Pain and Spine Specialists, Voorhees Township, New Jersey
  - Stony Brook University Medical Center, Stony Brook, New York
  - The Center for Clinical Research, LLC, Winston-Salem, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Neurospine Institute, Eugene, Oregon
  - Axis Spine Care, Tyler, Texas
  - Space City Pain Specialists, LLP, Webster, Texas
  - The Center for Pain Relief, Inc., Charleston, West Virginia
  - The Center for Pain relief Tri-State, Huntington, West Virginia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Percutaneous Lumbar Decompression | Lumbar Epidural Steroid Injection
Started | 122 | 16
Completed | 105 | 11
Not Completed | 17 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Percutaneous Lumbar Decompression | Lumbar Epidural Steroid Injection | Total
Number analyzed (Participants) | 122 | 16 | 138
Age, Continuous [Mean (Standard Deviation); unit: Years] | 72.9 (9.73) | 69.94 (9.73) | 72.56 (9.91)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 9 | 81
  Male | 50 | 7 | 57

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a 2-point Improvement in Visual Analogue Scale
Description: The primary endpoint for evaluating effectiveness will be the proportion of subjects in each group achieving at least a 2-point improvement from baseline in the Visual Analog Scale.
Time Frame: 16 weeks
Population: All participants who reported 16 week outcomes are included in this analysis.
Measure: Number; unit: percentage of responders
Arm/Group | Percutaneous Lumbar Decompression | Lumbar Epidural Steroid Injection
Number analyzed (Participants) | 114 | 13
percentage of responders | 65.71 | 46.15

ADVERSE EVENTS:
Arm/Group | Percutaneous Lumbar Decompression | Lumbar Epidural Steroid Injection
Serious Adverse Events (participants affected / at risk) | 4/122 | 2/16
Other Adverse Events (participants affected / at risk) | 8/122 | 0/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Percutaneous Lumbar Decompression (N=122) | Lumbar Epidural Steroid Injection (N=16)
FEVER (HOSPITALIZED) (Infections and infestations) | 1 (1) | 0 (0)
PROGRESSION OF SPINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
BRONCHITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1) | 0 (0)
PNEUMONIA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
CHEST PAIN (Cardiac disorders) | 0 (0) | 1 (1)
ORTHOSTASIS (Cardiac disorders) | 0 (0) | 1 (1)
SUBARACHNOID HEMORRHAGE (Vascular disorders) | 0 (0) | 1 (1)
SUBDURAL HEMATOMA (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Percutaneous Lumbar Decompression (N=122) | Lumbar Epidural Steroid Injection (N=16)
RIGHT BUTTOCK PAIN DUE TO TRANSFORAMINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Heart Block (Cardiac disorders) | 1 (1) | 0 (0)
RIGHT BUTTOCK PAIN DUE TO TRANSFORAMINAL STENOSIS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
UTI (Infections and infestations) | 1 (1) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
EXACERBATION OF LEG PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
INTERMITTENT LEFT SIDE SACROILLIAC PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
EXACERBATION OR RADICULAR PAIN RIGHT SIDE LEG (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No